CLINICAL TRIAL: NCT06682091
Title: Management and Outcome of Mesh Infections After Abdominoplasty in a Tertiary Care Center in France
Brief Title: Management and Outcome of Mesh Infection After Abdominoplasty in a Tertiary Care Centre
Acronym: MOCOMI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0567
Record Dates: First submitted 2024-06-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Abdominal Infection
Keywords: mesh infection; abdominoplasty
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of patients admitted for an abdominal mesh infection at Hospices Civils de Lyon: No intervention. Retrospective data collection.

SUMMARY:
Hernia repair is among most frequent surgical interventions. The use of abdominal mesh in hernia repair has become the Gold Standard strategy, reducing the risk of relapse.

The mesh infection risk is estimated lower than 1% in simple situations, but can increase up to 20% in complicated patients. Risk factors are well known, but we lack data regarding the therapeutic strategies and outcomes.

This study aims to describe the characteristics and management of abdominal mesh infections, and the related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* parietal mesh infection
* age > 18

Exclusion Criteria:

* Non French speaking patients.
* Persons under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects taken in care for abdominal mesh infection in the Hospices Civils de Lyon from 2010 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Treatment failure. | Retrospective analysis from initial treatment to any treatment failure within 2010 to 2023
  Clinical failure = persistance of the infection. Time of failure is the time of change of therapeutic strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse - Centre de reference des infection ostéo-articulaires de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No